CLINICAL TRIAL: NCT02562677
Title: Effect of TNS for Major Depressive Disorder in the Elderly: a Phase II Randomized Controlled Trial
Brief Title: TNS for Treating Major Depressive Disorder in the Elderly
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Santa Casa Medical School (Other)
Responsible Party: Principal Investigator, Pedro Shiozawa, Coordinator - Interdisciplinary Center for Clinical Neuromodulation, Santa Casa Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNS for Elderly
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Major Depressive Disorder; Elderly
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACTIVE tNS (Experimental): TNS will be applied by the external simulator (Monarch). The stimulation will be conducted at a frequency of 120 Hz with pulse duration of 250 microseconds. The current intensity will be individually established and should be equivalent to a slight feeling of not painful paresthesia .The stimulus generates a pulse and asymmetric biphasic waveform. Electrodes (25cm2) will be placed on the forehead just above the supraorbital foramen bilaterally. The study protocol will follow the rational of our previous trials with TNS.
  Interventions: Device: Transcutaneous Trigeminal Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Trigeminal Nerve Stimulation

SUMMARY:
This is a phase II, open-label clinical trial. This clinical trial has as primary objective to evaluate changes in EEG of a Trigeminal Nerve Stimulation (TNS) treatment protocol for elderly patients with moderate / severe depressive episode.

ELIGIBILITY:
Inclusion Criteria:

1. patients between 65 and 99 years
2. patients with a diagnosis of depression according to the SCID
3. score greater than or equal to 18 on the Hamilton Rating Scale 17-item version (equivalent to moderate or severe depressive episode)
4. agreement to participate in the study as recommended in the IC.

Exclusion Criteria:

1. patients with psychiatric indication for hospitalization
2. patients with psychiatric comorbidity
3. patients with a diagnosis of personality disorder
4. presence of severe neurological or medical diseases such as neoplasms in activity, neurodegenerative diseases and chronic diseases uncompensated.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depressive Rating Scale version 17 items (HDRS-17) | Change from baseline in depressive symptoms at 2 weeks ]
  This clinical trial has as primary objective to evaluate the effect of the Trigeminal Nerve Stimulation (TNS) on depressive symptoms measured by the Hamilton Depressive Rating Scale version 17 items (HDRS-17) in elderly patients with moderate / severe depressive episode

REFERENCES:
- [Result] Shiozawa P, Duailibi MS, da Silva ME, Cordeiro Q. Trigeminal nerve stimulation (TNS) protocol for treating major depression: an open-label proof-of-concept trial. Epilepsy Behav. 2014 Oct;39:6-9. doi: 10.1016/j.yebeh.2014.07.021. Epub 2014 Aug 23. PMID 25150403
- [Result] Shiozawa P, Silva ME, Carvalho TC, Cordeiro Q, Brunoni AR, Fregni F. Transcutaneous vagus and trigeminal nerve stimulation for neuropsychiatric disorders: a systematic review. Arq Neuropsiquiatr. 2014 Jul;72(7):542-7. doi: 10.1590/0004-282x20140061. PMID 25054988